CLINICAL TRIAL: NCT05765864
Title: Influences on and Prevention of Self-harm Behaviour Among the Most At-risk Adolescents
Brief Title: Self-harm Behaviour Among the Most At-risk Adolescents
Acronym: SH-MARA
Status: Recruiting | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Collaborators: University Medical Centre Ljubljana (Other); University Maribor (Other); University Psychiatric Clinic Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Drobnič Radobuljac, Assist. prof. Maja Drobnič Radobuljac, MD, PhD, University of Ljubljana, Faculty of Medicine
Other Study IDs: Adolescent self-harm
Record Dates: First submitted 2023-02-12; First posted 2023-03-13 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Self-harm; Personality Disorder, Borderline; Epigenetic Disorder; Non-Suicidal Self Injury; Change; Mental; Difference, Individual
Keywords: adolescent; deliberate self-harm; risk and protective factors; suicidal behavior; non-suicidal self-injury; risk assessment; attachment; genetics; epigenetics
MeSH Terms: conditions — Self-Injurious Behavior; Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The genomic DNA is going to be isolated according to the established laboratory protocol using FlexGene DNA kit (Qiagen Germany) and 5 mL EDTA-blood sample. Isolated DNA will be stored at 4°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: The Enrollment Kit and Time1 Kit will be administered at enrollment, Time2 Kit will be administered before discharge and Time 3 kit after 6 and 18 months post hospitalization (see Detailed description and Study Protocol). The interventions will be Treatment as usual.
  Interventions: Diagnostic Test: Enrollment questionnaire, General questionnaire1, General questionnaire2, General questionnaire3; Diagnostic Test: Columbia Suicide Severity Rating Scale (CSSRS); Diagnostic Test: The Brief Non-Suicidal Self-Injury Assessment Tool (B-NSSI-AT); Diagnostic Test: Experiences in Close Relationships-Relationship Structures (ECR-RS); Diagnostic Test: Trauma Symptom Checklist for Children (TSCC); Diagnostic Test: Personality Assessment Inventory-Adolescent (PAI-A); Diagnostic Test: Inventory Of Statements About Self-Injury; ISAS; Diagnostic Test: The Level of Personality Functioning Scale-Brief Form 2.0; LPFSBF 2.0; Diagnostic Test: Borderline Personality Features Scale, BPFSC-11; Other: Dynamic Appraisal of Situational Aggression-Youth Version (DASA-YV); Other: Adolescent Self-Harm Risk Scale; ASHRS; Diagnostic Test: Lifetime Incidence of Traumatic Events questionnaire (LITE); Genetic: Genetic methods
- Controls: The Enrollment Kit and the Time Kit1 will be administered (see Detailed description and Study Protocol).
  Interventions: Diagnostic Test: Enrollment questionnaire, General questionnaire1, General questionnaire2, General questionnaire3; Diagnostic Test: Columbia Suicide Severity Rating Scale (CSSRS); Diagnostic Test: The Brief Non-Suicidal Self-Injury Assessment Tool (B-NSSI-AT); Diagnostic Test: Experiences in Close Relationships-Relationship Structures (ECR-RS); Diagnostic Test: Trauma Symptom Checklist for Children (TSCC); Diagnostic Test: Personality Assessment Inventory-Adolescent (PAI-A); Diagnostic Test: Inventory Of Statements About Self-Injury; ISAS; Diagnostic Test: The Level of Personality Functioning Scale-Brief Form 2.0; LPFSBF 2.0; Diagnostic Test: Borderline Personality Features Scale, BPFSC-11; Other: Dynamic Appraisal of Situational Aggression-Youth Version (DASA-YV); Other: Adolescent Self-Harm Risk Scale; ASHRS; Diagnostic Test: Lifetime Incidence of Traumatic Events questionnaire (LITE); Genetic: Genetic methods

INTERVENTIONS:
Diagnostic Test: Enrollment questionnaire, General questionnaire1, General questionnaire2, General questionnaire3 — The questionnaires will cover general and demographic data, information on previous treatments, medication received, mental disorder at discharge (ICD), psychosocial situations (ICD), physical illnesses (ICD), COVID status (vaccinated, recovered, tested), use of psychoactive substances, history of self-harm, suicide attempts, school performance, experience with peers, sexual orientation and identity, residence, family composition, family history of mental disorders, self-harm and suicide attempts.
Diagnostic Test: Columbia Suicide Severity Rating Scale (CSSRS) — The questionnaire is scientifically supported, has the most evidence of utility and efficacy, and is internationally accepted. It has been translated into more than 100 different languages, including Slovene. It is easy to use, suitable for all age groups and adapted for successful use outside the hospital setting, for example in schools, colleges, police, military and elsewhere. It contains 2 screening questions on suicidality and 4 more specific questions, 6 items in total.
  Posner K, Brown GK, Stanley B, et al. Am J Psychiatry 2011;168:1266-77.
Diagnostic Test: The Brief Non-Suicidal Self-Injury Assessment Tool (B-NSSI-AT) — used for research purposes to assess the core characteristics of NSSI (form, frequency, function) as well as the secondary characteristics of NSSI (habituation, context of NSSI, perceived impact on life and treatment).
  Whitlock J, Exner-Cortens D, Purington A. Psychol Assess 2014;26:935-46.
Diagnostic Test: Experiences in Close Relationships-Relationship Structures (ECR-RS) — Assesses the pattern of attachment to attachment figures (friend, romantic partner, mother, father) in adults and adolescents. The questionnaire has been officially translated into Slovene and used with several samples of Slovene adults and adolescents.
  Fraley RC, Waller NG, Brennan KA. J Pers Soc Psychol 2000;78:350-65.
Diagnostic Test: Trauma Symptom Checklist for Children (TSCC) — The questionnaire helps to assess children's/adolescents' experiences of various traumatic experiences, such as physical or sexual violence, peer violence, loss, witnessing violent acts, natural disasters, etc. The questionnaire consists of 6 clinical scales (Anxiety, Depression, Anger, Post-traumatic Stress Symptom, Dissociativeness (two subscales), Sexual Concerns) and 2 validity scales. 6 clinical scales (Anxiety, Depressiveness, Anger, Post-traumatic Stress Symptom, Dissociativeness (two subscales), and 2 validity scales) are included.
  https://www.center-pds.si/Katalogtestov/Kliničnitesti/Vprašalnikotravmatiziranostiotrokinmladostnik. aspx
Diagnostic Test: Personality Assessment Inventory-Adolescent (PAI-A) — An objective-type self-assessment questionnaire for assessing personality in adolescents. It has 264 items to be answered on a 4-point scale. 22 independent scales are obtained (Inconsistency, Rarity, Negative impression, Positive impression, Physical complaints, Anxiety, Anxiety-related disorders, Depressiveness, Mania, Paranoid, Schizophrenia, Borderline traits, Antisocial traits, Alcohol problems, Drug problems, Aggressiveness, Suicidal ideation, Stress, Lack of support, Refusal to deal, Dominance, Warmth).
  https://www.center-pds.si/Katalogtestov/Kliničnitesti/Vprašalnikzaocenoosebnosti-oblikazamladostnike-PAI-A.aspx
Diagnostic Test: Inventory Of Statements About Self-Injury; ISAS — A self-assessment questionnaire used for research purposes to assess the basic characteristics of NSSI (form, frequency, function, time to event). It also assesses the desire to stop. The questionnaire has been previously translated into Slovene and used in a population of adolescents with self-injurious behaviour.
  Glenn CR, Klonsky ED. One-year test-retest reliability of the Inventory of Statements about Self-Injury (ISAS). Assessment. 2011 Sep;18(3):375-8. doi: 10.1177/1073191111411669.
Diagnostic Test: The Level of Personality Functioning Scale-Brief Form 2.0; LPFSBF 2.0 — A short, user-friendly instrument that gives a quick impression of the expression of personality pathology. It consists of 12 items grouped into two higher-order domains: self-functioning and interpersonal functioning. Participants are asked to rate the 12 items on a four-point Likert scale ranging from 1 (completely false) to 4 (completely true). A total score (sum of all items), a self-functioning score (sum of items 1-6) and an interpersonal functioning score (sum of items 7-12) can be calculated. Satisfactory internal consistency and promising construct validity have been demonstrated. Sensitivity to change after three months of treatment was high.
  Weekers LC, Hutsebaut J, Kamphuis JH. The Level of Personality Functioning Scale-Brief Form 2.0: Update of a brief instrument for assessing level of personality functioning. Personal Ment Health 2019;13:3-14.
Diagnostic Test: Borderline Personality Features Scale, BPFSC-11 — The BPFS-C-11 includes BPD indicators such as affective instability, identity problems and negative attitudes. Responses to the items are on a 5-point Likert scale ranging from 'not at all true' to 'always true'. Studies have shown construct validity of interpretations of BPFS-C-11 scores through positive associations with other measures of BPD and positive associations with measures of BPD correlates, including emotional dysregulation. In a recent sample, the Cronbach's α over 4 years of follow-up was 0.86, 0.85, 0.86 and 0.90, respectively. The scale has been officially translated into Slovenian and will be used with the permission of the authors. It is intended for use by children and adolescents aged 9-11 years and consists of 11 items.
  Sharp, C., Steinberg, L., Temple, J., Newlin, E. An 11-Item Measure to Assess Borderline Traits in Adolescents: Refinement of the BPFSC Using IRT . Personality Disorders: Theory, Research, and Treatment 2014;5(1):70-78.
Other: Dynamic Appraisal of Situational Aggression-Youth Version (DASA-YV) — It's a professional assessment tool which provides a daily assessment of the risk of heteroaggression. The evaluation is efficient and takes less than five minutes. The nurse in charge of each patient completes the DASA-YV once a day.
  Dutch SG, Patil N. Validating a Measurement Tool to Predict Aggressive Behavior in Hospitalized Youth. J Am Psychiatr Nurses Assoc 2019;25:396-404.
Other: Adolescent Self-Harm Risk Scale; ASHRS — It's a professional assessment tool which provides a daily assessment of the risk of heteroaggression. This is the scale we developed for the present study. It will be used to assess and predict the short-term risk of self-harm behaviour during hospitalisation (assessment at admission) and the long-term risk after discharge (assessment at discharge).
Diagnostic Test: Lifetime Incidence of Traumatic Events questionnaire (LITE) — Is a short checklist for screening and assessing the exposure to trauma in children and adolescents. It covers a broad range of potentially upsetting situations that can cause trauma to children and adolescents, such as a car accident, fire, death of a family member, exposure to threats, sexual assault, or witnessing violence. The questionnaire had been validated on a Slovene population of children and adolesscents.
  Greenwald R, Rubin A. Assessment of posttraumatic symptoms in children:
  development and preliminary validation of parent and child scales. Res Soc Work Pract. (1999) 9:61-75. doi: 10.1177/104973159900900105 Uršicˇ K, Bucik V, Klemencˇ icˇ S, Bratina N, Battelino T, Dovcˇ K and Drobnicˇ Radobuljac M (2021) Validation of the Lifetime Incidence of Traumatic Events (LITE-S/P) Questionnaires in Children and Adolescents in Slovenia. Front. Psychiatry 12:665315. doi: 10.3389/fpsyt.2021.665315
Genetic: Genetic methods — DNA isolation, Sequencing, Libraries preparation, Analisys; Bioinformatics (Base Calling, Variant Calling, Quantification and evaluation of short tandem repetitions, Methylation sites detection).

SUMMARY:
In the proposed study, three objectives will be pursued:

1. To develop a method to identify more effectively the acute and long-term risk of adolescents with the most threatening self-harm behaviours.
2. To identify the factors that influence the risk of self-harm behaviours and the success of treatment/treatment of these behaviours in the most at-risk adolescents (changes in these factors).
3. Develop guidelines for more effective treatment of the most at-risk adolescents.

For this purpose, a sample of approximately 200 young people who will be hospitalised for suicide risk (the most at risk in Slovenia) and an approximately equal number of healthy adolescents will be included. At inclusion, the presence of several factors will be assessed by reviewing demographic data, clinical diagnosis, self-assessment questionnaires and clinical psychological tests (CSSRS, B-NSSI-AT, ISAS, LPFS-BF2.0, BPFSC-11, TSCC, PAI, ECR-RS, DASA-YV, ASHRS), social assessment, and blood sampling for genetic analyses (DNA isolation, sequencing, nucleotide sequence recognition, quantification and evaluation of short tandem repeats, identification of methylation sites). Longitudinal tracking of autoaggressive events and heteroaggressive events during hospitalisation will be performed and recorded on an ongoing basis. The risk and protective factors of the adolescents most at risk will be compared with a control group of adolescents. The same factors will be reassessed in the most at-risk adolescents after 6 and 18 months of treatment as usual. The data will be collected in a data entry and storage system that will ensure the privacy of the data entered in accordance with the GDPR.

This will allow the investigators to identify young people at particular risk of severe self-harm behaviour more reliably, to target them for more intensive and effective treatment, and thus to improve their safety, quality of life and prognosis in the short and long term.

DETAILED DESCRIPTION:
DESCRIPTION OF THE RESEARCH PROJECT "Influences on and prevention of self-harm behaviour among the most at-risk adolescents".

1. Scientific background Detailed in the attached Study Protocol
2. Detailed description of the work programme 2.1. Content and work programme The study will include a sample of approximately 200 young people who will be hospitalised for suicide risk (the most at risk in Slovenia) and an approximately equal number of healthy adolescents. At enrolment, the investigators will assess the presence of several factors by reviewing demographic data, clinical diagnosis, self-assessment questionnaires, social assessment, clinical psychological tests, rating scales and blood sampling for genetic analyses. They will longitudinally track autoaggressive events and heteroaggressive events in the patients during hospitalisation and keep a running record of them. The risk and protective factors of the most at-risk adolescents will be compared to a control group of healthy adolescents. The same factors in the most at-risk adolescents will be reassessed after 6 and 18 months of treatment. A detailed description of the study design is given in Figure 2 and Table 2 of Study Protocol.

2.2. Subjects: Subjects with inclusion and exclusion criteria are described in Table 2 (Study Protocol, WP2).

2.3. Methods: 2.3.1. Questionnaires and psychodiagnostic tools:

1. Enrollment questionnaire, General questionnaire1, General questionnaire2, General questionnaire3: The questionnaires will cover general and demographic data, information on previous treatments, medication received, mental disorder at discharge (ICD), psychosocial situations (ICD), physical illnesses (ICD), COVID status (vaccinated, recovered, tested), use of psychoactive substances, history of self-harm, suicide attempts, school performance, experience with peers, sexual orientation and identity, residence, family composition, family history of mental disorders, self-harm and suicide attempts.
2. Columbia Suicide Severity Rating Scale (CSSRS).
3. The Brief Non-Suicidal Self-Injury Assessment Tool (B-NSSI-AT).
4. Personality Assessment Inventory-Adolescent (PAI-A).
5. Trauma Symptom Checklist for Children (TSCC).
6. Experiences in Close Relationships-Relationship Structures (ECR-RS).
7. Dynamic Appraisal of Situational Aggression-Youth Version (DASA-YV).
8. Adolescent Self-Harm Risk Scale (ASHRS): this is the scale we developed for the present study.
9. The Level of Personality Functioning Scale-Brief Form 2.0 (LPFSBF 2.0).
10. Lifetime Incidence of Traumatic Events questionnaire (LITE).
11. Borderline Personality Features Scale (BPFSC-11).
12. Inventory Of Statements About Self-Injury (ISAS).

2.3.2. Genetic methods: DNA isolation: The genomic DNA is going to be isolated according to the established laboratory protocol using FlexGene DNA kit (Qiagen Germany) and 5 mL EDTA-blood sample. Isolated DNA will be stored at 4°C.

Sequencing: Sequencing will be performed on available in-house long-read sequencing technology nanopore PromethION (Oxford Nanopore Technologies). The ability to detect DNA modifications via differences in the electric current intensity produced from a nanopore read of an unmodified base and that of a modified base, enables the detection of DNA methylation in different CpGs from human natural DNA at epigenome-wide level.

Libraries will be prepared using ligation sequencing kit (SQK-LSK 109, Oxford Nanopore Technologies) in following stages: 1. NEBNext Ultra II End repair / dA-tailing, 2. ligation of the native barcodes, 3. ligation of sequencing adapters, 4. flow cell priming and DNA library loading (Flow Cell Priming Kit, Oxford Nanopore Technologies).

The analysis will be conducted using barcoded participants' DNA, enabling the simultaneous analysis of multiple participant's, by pooling the equimolar amount of DNA into a single pool, based on the observation groups. The sample pooling will reduce the effect of individual epigenome variability and enrich the cohort-specific epigenetic signals, potentially associated with the clinical phenotype.

Bioinformatics Base Calling: From the raw sequencing signal, the nucleotide sequences will be determined using the software tool Guppy, which is based on a predictive neural network model. The identified reads and their reliability will be stored in FASTQ files. For subsequent alignments of long reads, the human genome (GRCh38) will be used as a reference.

Variant Calling: Megalodon software (Oxford Nanopore Technologies) will be utilized for determining nucleotide sequences from the raw signal, alignment of readings on human reference genome and variant calling. The reliability of the findings will be additionally confirmed using the software tool Medaka (Oxford Nanopore Technologies). The tool uses a neural network model to identify genetic variants, based on constructed consensus sequences. Variant data will be stored in VCF files.

Quantification and evaluation of short tandem repetitions: Tandem-genotypes and STRique will be used to detect changes in length of tandem repeats, from aligned long DNA reads. In addition to the aligned reads input, the software tool STRique accepts the raw sequencing signal, based on which a hidden Markov model quantifies and evaluates the likelihood of a change. The validated changes in length of tandem repeats will be stored in TSV files.

Methylation sites detection: Different methylation-calling tools will be utilized using the METEORE software tool. The reliability of the methylated CpG islands found in the results will be demonstrated by the prediction models (random forest and multiple linear regression). Additionally, the detected methylated sites will be compared with the results of the Remora software (Oxford Nanopore Technologies). The locations of reliable methylation sites will be stored in BED and TSV files.

2.4. Conduct of the research "Influences on and prevention of self-harm behaviour among the most at-risk adolescents" The detailed survey process is described in Figure 2 and Table 2 of Study Protocol.

Detailed definition of the work packages of the research "Influences on and prevention of self-harm behaviour among the most at-risk adolescents".

2.4.1. WP 1: Establishment of a working research module on "Influences on and prevention of self-harm behaviour among the most at-risk adolescents".

Lead organisation: University of Ljubljana, Faculty of Medicine and Centre for Mental Health, University Psychiatric Clinic Ljubljana (UPKL) Participating organisations: the Clinical Institute of Special Laboratory Diagnostics of the Paediatric Clinic of the UKC Ljubljana (KISLD) and the Faculty of Electrical Engineering, Computer Science and Informatics of the University of Maribor (FERI) T1: At this stage, all questionnaires were prepared in sets with the corresponding survey numbers.

1. Enrollment kit (Screening questionnaire, CSSRS, B-NSSI-AT)
2. Time1 kit (General Questionnaire1, PAI-A, TSCC, ECR-RS, DASA-YV, ASHRS, LPFSBF 2.0, LITE, BPFSC-11, ISAS), venous blood sample collection for genetic analyses
3. Time2 kit (DASA-YV tracing, Incident Report (commited and prevented), General Questionnaire2)
4. Time3 kit (General Questionnaire3, CSSRS, B-NSSI-AT, PAI-A subscales, TSCC subscales, ECR-RS, DASA-YV, ASHRS, LPFSBF 2.0, LITE, BPFSC-11), venous blood sample collection for genetic analyses.

T2: Development of a protocol for subject enrolment and data acquisition, storage and analysis. This work included the preparation of information materials for subjects and parents/guardians, informed consents/assents and a detailed protocol that will be accessible to the investigators throughout the study.

T3: Preparation of the data entry and storage system: The data entry and storage information system will be prepared so that it will enable data entry via pre-prepared templates for initial and intermediate reporting of measurements. The system will ensure data privacy, as access will be restricted to anonymized data and allowed only for the purposes of analysis (in line with the General Data Protection Regulation (EU) 2016/679 (GDPR)). The system will ensure that data is safely deleted after the project is completed (according to the GDPR). The information system will be physically located in the Republic of Slovenia, and physical access to the hardware will be limited only to administrative activities by qualified personnel.

T4: Education and training of the working group: This part will consist of several educational sessions for the different members of the working group: a. Patient involvement, involvement of pupils and students of the control group (assessment of the fulfilment of inclusion/exclusion criteria, information about the study, obtaining consent from adolescents and relatives), b. Collection of questionnaire responses, c. Collection of biological samples, d. Data collection during hospitalisation, e. Follow-up. Initial training sessions will be followed by more frequent follow-up of the study processess, possible complications, necessary adjustments of the protocol according to the initial experience (project manager Maja Drobnič Radobuljac) and re-training if necessary.

2.4.2. WP 2: Study and control group recruitment, data collection, patient follow-up.

Lead organisation: UPKL Participating organisations: KISLD and FERI

Objectives:

In this work package the investigators will focus on the involvement of patients and healthy adolescents. The work package includes capturing all patient data at Time 1 and tracking patients during hospitalization until discharge (Time 2) and recapturing data at Time 3 (Figure 2 of Study Protocol). On the control group side, only data at Time 1 will be captured (Figure 2 of Study Protocol). This work package has three main objectives: enrollment of hospitalized and healthy adolescents, data collection and follow-up.

Tasks:

T1: Enrollment of hospitalised adolescents. The Enrollment Kit and the Time1 Kit will be administered (see Figure 2 of Study Protocol), and the Time2 Kit will be administered during hospitalisation and at discharge.

T2: Enrollment of healthy adolescents (control group). The Enrollment Kit and the Time Kit1 will be administered (see Figure 2 of Study Protocol).

T3: Data collection. Data from hospitalised patients will be collected by administering the Enrollment, Time1, Time2 kits (see Figure 2 of Study Protocol). Adolescents in the control group will have the Enrollment and Time1 kits administered immediately on enrollment, no other data will be collected from these adolescents (see Figure 2 of Study Protocol). In the event that any of the adolescents approached appeared to be in need of help for self-injurious behaviour or other overt mental disorders, they will be referred for appropriate treatment.

T4: Tracking. Six and 18 months after the end of the hospitalization, the investigators will contact the patients again and administer the Time3 kit (see Figure 2 of Study Protocol). If any of the adolescents approached appear to need help for self-injurious behaviour or other overt mental disorders, they will be referred for appropriate treatment.

2.4.3. WP 3: Analysis of extracted materials, data entry and statistical analysis Lead organisation: UPKL, KISLD and FERI Participating organisations: UPKL, KISLD and FERI

Objectives:

The first objective is to identify the factors influencing the occurrence of the most threatening forms of self-injurious behaviour in adolescents.

The second aim is to assess the factors that influence change in risk of self-harm behaviour in the most at-risk adolescents.

The third objective is to develop an instrument (scale) for rapid assessment of short- and medium-term risk of self-harm in adolescents (ASHRS).

The details are in the Study Protocol.

ELIGIBILITY:
CLINICAL GROUP:

Inclusion Criteria:

* Suicidality
* Self-harming with no intention to die

Exclusion Criteria:

* Confirmed acute psychotic disorder
* Intellectual disability
* Severe physical illness (e.g. cardiovascular or renal disease)
* Disease of the central nervous system (e.g. encephalitis, brain injury or haemorrhage, epilepsy)
* Acute poisoning (including with psychoactive substances)

CONTROL GROUP:

Inclusion Criteria:

- Age 13-19

Exclusion criteria:

* Suicidality
* Self-harming with no intention to die
* Known mental disorder (e.g. depression, bipolar disorder, schizophrenia, intellectual disability)
* Severe physical illness (e.g. cardiovascular or renal disease)
* Disease of the central nervous system (e.g. encephalitis, brain injury or haemorrhage, epilepsy)
* Acute poisoning (including with psychoactive substances)
* Mental disorder, history of suicidality or self-injurious behaviour in a first-degree relative (a parent or a sibling).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: CLINICAL GROUP:
  * patients hospitalized in the Intensive Child and Adolescent Psychiatry Unit or the Unit for Adolescent Psychiatry of the Centre for Mental Health University Psychiatric Clinic Ljubljana
  * aged between 13 and 19 years.
  * In the case of consent, parents will also be asked for consent for those under 15 years of age.
  CONTROL GROUP:
  * 8th grade students in primary school,
  * 1st year students in secondary school
  * 1st year students in college
  * aged 13-19 years
  * Attending a regular systematic review. These scheduled regular systematic examinations are accompanied by venous blood sampling.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Self-harm incident | "through study completion, an average of 1 year"
  Registered incident of self-harm
Prevented self-harm incident | "up to 12 weeks"
  Registration of an intended self-harm prevented by hospital staff (nurses)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Drobnič Radobuljac, Principal Investigator — University Psychiatric Clinic Ljubljana
Locations (2):
- Slovenia (2):
  - Medical Faculty - University of Ljubljana, Ljubljana
  - University Psychiatric Clinic Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giedd JN, Blumenthal J, Jeffries NO, Castellanos FX, Liu H, Zijdenbos A, Paus T, Evans AC, Rapoport JL. Brain development during childhood and adolescence: a longitudinal MRI study. Nat Neurosci. 1999 Oct;2(10):861-3. doi: 10.1038/13158. No abstract available. PMID 10491603
- [Background] Spear LP. Adolescent neurodevelopment. J Adolesc Health. 2013 Feb;52(2 Suppl 2):S7-13. doi: 10.1016/j.jadohealth.2012.05.006. PMID 23332574
- [Background] Steinberg L, Morris AS. Adolescent development. Annu Rev Psychol. 2001;52:83-110. doi: 10.1146/annurev.psych.52.1.83. PMID 11148300
- [Background] Stoep AV, McCauley E, Flynn C, Stone A. Thoughts of death and suicide in early adolescence. Suicide Life Threat Behav. 2009 Dec;39(6):599-613. doi: 10.1521/suli.2009.39.6.599. PMID 20121323
- [Background] Radobuljac MD, Bratina NU, Battelino T, Tomori M. Lifetime prevalence of suicidal and self-injurious behaviors in a representative cohort of Slovenian adolescents with type 1 diabetes. Pediatr Diabetes. 2009 Nov;10(7):424-31. doi: 10.1111/j.1399-5448.2009.00501.x. Epub 2009 Apr 8. PMID 19490494
- [Background] Bridge JA, Goldstein TR, Brent DA. Adolescent suicide and suicidal behavior. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):372-94. doi: 10.1111/j.1469-7610.2006.01615.x. PMID 16492264
- [Background] SURS. Slovenija: Statistični Urad Republike Slovenije; 2021.
- [Background] Wilkinson P, Goodyer I. Non-suicidal self-injury. Eur Child Adolesc Psychiatry. 2011 Feb;20(2):103-8. doi: 10.1007/s00787-010-0156-y. Epub 2011 Jan 11. PMID 21222215
- [Background] Surveillance report 2016 - Self-harm in over 8s: short-term management and prevention of recurrence (2004) NICE guideline CG16 and Self-harm in over 8s: long term management (2011) NICE guideline CG133 [Internet]. London: National Institute for Health and Care Excellence (NICE); 2016 Sep 30. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK552073/ PMID 31891461
- [Background] Diagnostic and Statistical Manual of Mental Disorders. Fifth Edition ed. Arlington, VA: American Psychiatric Association; 2013.
- [Background] Favazza AR, Conterio K. Female habitual self-mutilators. Acta Psychiatr Scand. 1989 Mar;79(3):283-9. doi: 10.1111/j.1600-0447.1989.tb10259.x. PMID 2711856
- [Background] Favazza AR. Nonsuicidal self-injury: How categorization guides treatment. Current Psychiatry 2012;11(3):21-5.
- [Background] Tomori M, Zalar B, Plesnicar BK. Gender differences in psychosocial risk factors among Slovenian adolescents. Adolescence. 2000 Autumn;35(139):431-43. PMID 11130589
- [Background] Žerjav Ž, Drobnič Radobuljac M. Medicinski Razgledi 2019;58:417-27.
- [Background] Kiric B, Leben Novak L, Lusicky P, Drobnic Radobuljac M. Suicidal Behavior in Emergency Child and Adolescent Psychiatric Service Users Before and During the 16 Months of the COVID-19 Pandemic. Front Psychiatry. 2022 May 11;13:893040. doi: 10.3389/fpsyt.2022.893040. eCollection 2022. PMID 35633784
- [Background] Swannell SV, Martin GE, Page A, Hasking P, St John NJ. Prevalence of nonsuicidal self-injury in nonclinical samples: systematic review, meta-analysis and meta-regression. Suicide Life Threat Behav. 2014 Jun;44(3):273-303. doi: 10.1111/sltb.12070. Epub 2014 Jan 15. PMID 24422986
- [Background] Plener PL, Allroggen M, Kapusta ND, Brahler E, Fegert JM, Groschwitz RC. The prevalence of Nonsuicidal Self-Injury (NSSI) in a representative sample of the German population. BMC Psychiatry. 2016 Oct 19;16(1):353. doi: 10.1186/s12888-016-1060-x. PMID 27760537
- [Background] Groschwitz RC, Plener PL, Kaess M, Schumacher T, Stoehr R, Boege I. The situation of former adolescent self-injurers as young adults: a follow-up study. BMC Psychiatry. 2015 Jul 18;15:160. doi: 10.1186/s12888-015-0555-1. PMID 26187150
- [Background] Kaess M, Parzer P, Mattern M, Plener PL, Bifulco A, Resch F, Brunner R. Adverse childhood experiences and their impact on frequency, severity, and the individual function of nonsuicidal self-injury in youth. Psychiatry Res. 2013 Apr 30;206(2-3):265-72. doi: 10.1016/j.psychres.2012.10.012. Epub 2012 Nov 16. PMID 23159195
- [Background] Zahl DL, Hawton K. Repetition of deliberate self-harm and subsequent suicide risk: long-term follow-up study of 11,583 patients. Br J Psychiatry. 2004 Jul;185:70-5. doi: 10.1192/bjp.185.1.70. PMID 15231558
- [Background] Moran P, Coffey C, Romaniuk H, Olsson C, Borschmann R, Carlin JB, Patton GC. The natural history of self-harm from adolescence to young adulthood: a population-based cohort study. Lancet. 2012 Jan 21;379(9812):236-43. doi: 10.1016/S0140-6736(11)61141-0. Epub 2011 Nov 16. PMID 22100201
- [Background] Carballo JJ, Llorente C, Kehrmann L, Flamarique I, Zuddas A, Purper-Ouakil D, Hoekstra PJ, Coghill D, Schulze UME, Dittmann RW, Buitelaar JK, Castro-Fornieles J, Lievesley K, Santosh P, Arango C; STOP Consortium. Psychosocial risk factors for suicidality in children and adolescents. Eur Child Adolesc Psychiatry. 2020 Jun;29(6):759-776. doi: 10.1007/s00787-018-01270-9. Epub 2019 Jan 25. PMID 30684089
- [Background] Beautrais AL, Collings SCD, Ehrhardt P, K H. Suicide Prevention - A review of evidence of risk and protective factors, and points of effective intervention. In: Health Mo, ed. Wellington, NZ2005.
- [Background] Goldston DB, Daniel SS, Reboussin DM, Reboussin BA, Frazier PH, Kelley AE. Suicide attempts among formerly hospitalized adolescents: a prospective naturalistic study of risk during the first 5 years after discharge. J Am Acad Child Adolesc Psychiatry. 1999 Jun;38(6):660-71. doi: 10.1097/00004583-199906000-00012. PMID 10361783
- [Background] Clarke S, Allerhand LA, Berk MS. Recent advances in understanding and managing self-harm in adolescents. F1000Res. 2019 Oct 24;8:F1000 Faculty Rev-1794. doi: 10.12688/f1000research.19868.1. eCollection 2019. PMID 31681470
- [Background] Chung DT, Ryan CJ, Hadzi-Pavlovic D, Singh SP, Stanton C, Large MM. Suicide Rates After Discharge From Psychiatric Facilities: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Jul 1;74(7):694-702. doi: 10.1001/jamapsychiatry.2017.1044. PMID 28564699
- [Background] Hawton K, Bergen H, Cooper J, Turnbull P, Waters K, Ness J, Kapur N. Suicide following self-harm: findings from the Multicentre Study of self-harm in England, 2000-2012. J Affect Disord. 2015 Apr 1;175:147-51. doi: 10.1016/j.jad.2014.12.062. Epub 2015 Jan 8. PMID 25617686
- [Background] Hawton K, Bale L, Brand F, Townsend E, Ness J, Waters K, Clements C, Kapur N, Geulayov G. Mortality in children and adolescents following presentation to hospital after non-fatal self-harm in the Multicentre Study of Self-harm: a prospective observational cohort study. Lancet Child Adolesc Health. 2020 Feb;4(2):111-120. doi: 10.1016/S2352-4642(19)30373-6. Epub 2020 Jan 8. PMID 31926769
- [Background] King CA, Grupp-Phelan J, Brent D, Dean JM, Webb M, Bridge JA, Spirito A, Chernick LS, Mahabee-Gittens EM, Mistry RD, Rea M, Keller A, Rogers A, Shenoi R, Cwik M, Busby DR, Casper TC; Pediatric Emergency Care Applied Research Network. Predicting 3-month risk for adolescent suicide attempts among pediatric emergency department patients. J Child Psychol Psychiatry. 2019 Oct;60(10):1055-1064. doi: 10.1111/jcpp.13087. Epub 2019 Jul 21. PMID 31328282
- [Background] Bjureberg J, Ohlis A, Ljotsson B, D'Onofrio BM, Hedman-Lagerlof E, Jokinen J, Sahlin H, Lichtenstein P, Cederlof M, Hellner C. Adolescent self-harm with and without suicidality: cross-sectional and longitudinal analyses of a Swedish regional register. J Child Psychol Psychiatry. 2019 Mar;60(3):295-304. doi: 10.1111/jcpp.12967. Epub 2018 Sep 12. PMID 30207392
- [Background] Brent DA, Baugher M, Bridge J, Chen T, Chiappetta L. Age- and sex-related risk factors for adolescent suicide. J Am Acad Child Adolesc Psychiatry. 1999 Dec;38(12):1497-505. doi: 10.1097/00004583-199912000-00010. PMID 10596249
- [Background] Olfson M, Shaffer D, Marcus SC, Greenberg T. Relationship between antidepressant medication treatment and suicide in adolescents. Arch Gen Psychiatry. 2003 Oct;60(10):978-82. doi: 10.1001/archpsyc.60.9.978. PMID 14557142
- [Background] Tomori M, Zalar B. Gender differences among adolescent suicide attempters and nonattempters. Int J Adolesc Med Health. 2011 May 20;12(2-3):177-90. doi: 10.1515/IJAMH.2000.12.2-3.177. No abstract available. PMID 22912289
- [Background] Wichstrom L, Hegna K. Sexual orientation and suicide attempt: a longitudinal study of the general Norwegian adolescent population. J Abnorm Psychol. 2003 Feb;112(1):144-51. PMID 12653422
- [Background] Brent DA, Mann JJ. Family genetic studies, suicide, and suicidal behavior. Am J Med Genet C Semin Med Genet. 2005 Feb 15;133C(1):13-24. doi: 10.1002/ajmg.c.30042. PMID 15648081
- [Background] Zalsman G, Frisch A, Bromberg M, Gelernter J, Michaelovsky E, Campino A, Erlich Z, Tyano S, Apter A, Weizman A. Family-based association study of serotonin transporter promoter in suicidal adolescents: no association with suicidality but possible role in violence traits. Am J Med Genet. 2001 Apr 8;105(3):239-45. doi: 10.1002/ajmg.1261. PMID 11353442
- [Background] Zalsman G, Frisch A, King RA, Pauls DL, Grice DE, Gelernter J, Alsobrook J, Michaelovsky E, Apter A, Tyano S, Weizman A, Leckman JF. Case control and family-based studies of tryptophan hydroxylase gene A218C polymorphism and suicidality in adolescents. Am J Med Genet. 2001 Jul 8;105(5):451-7. doi: 10.1002/ajmg.1406. PMID 11449398
- [Background] Brent DA, Melhem N. Familial transmission of suicidal behavior. Psychiatr Clin North Am. 2008 Jun;31(2):157-77. doi: 10.1016/j.psc.2008.02.001. PMID 18439442
- [Background] McGirr A, Turecki G. The relationship of impulsive aggressiveness to suicidality and other depression-linked behaviors. Curr Psychiatry Rep. 2007 Dec;9(6):460-6. doi: 10.1007/s11920-007-0062-2. PMID 18221625
- [Background] Jang KL, Livesley WJ, Vernon PA, Jackson DN. Heritability of personality disorder traits: a twin study. Acta Psychiatr Scand. 1996 Dec;94(6):438-44. doi: 10.1111/j.1600-0447.1996.tb09887.x. PMID 9020996
- [Background] Maciejewski DF, Creemers HE, Lynskey MT, Madden PA, Heath AC, Statham DJ, Martin NG, Verweij KJ. Overlapping genetic and environmental influences on nonsuicidal self-injury and suicidal ideation: different outcomes, same etiology? JAMA Psychiatry. 2014 Jun;71(6):699-705. doi: 10.1001/jamapsychiatry.2014.89. PMID 24760386
- [Background] Gorodetsky E, Carli V, Sarchiapone M, Roy A, Goldman D, Enoch MA. Predictors for self-directed aggression in Italian prisoners include externalizing behaviors, childhood trauma and the serotonin transporter gene polymorphism 5-HTTLPR. Genes Brain Behav. 2016 Jun;15(5):465-73. doi: 10.1111/gbb.12293. Epub 2016 May 5. PMID 27062586
- [Background] Dell'osso L, Mandelli L, Carlini M, Bouanani S, Rotondo A, Conversano C, Serretti A, Marazziti D. Temperamental and genetic predictors of suicide attempt and self-mutilation. Neuropsychobiology. 2013;68(4):250-7. doi: 10.1159/000356228. Epub 2013 Nov 21. PMID 24280759
- [Background] Steiger H, Fichter M, Bruce KR, Joober R, Badawi G, Richardson J, Groleau P, Ramos C, Israel M, Bondy B, Quadflieg N, Bachetzky N. Molecular-genetic correlates of self-harming behaviors in eating-disordered women: findings from a combined Canadian-German sample. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jan 15;35(1):102-6. doi: 10.1016/j.pnpbp.2010.09.012. Epub 2010 Sep 29. PMID 20869421
- [Background] Bernegger A, Kienesberger K, Carlberg L, Swoboda P, Ludwig B, Koller R, Inaner M, Zotter M, Kapusta N, Aigner M, Haslacher H, Kasper S, Schosser A. The Impact of COMT and Childhood Maltreatment on Suicidal Behaviour in Affective Disorders. Sci Rep. 2018 Jan 12;8(1):692. doi: 10.1038/s41598-017-19040-z. PMID 29330410
- [Background] Joyce PR, McKenzie JM, Mulder RT, Luty SE, Sullivan PF, Miller AL, Kennedy MA. Genetic, developmental and personality correlates of self-mutilation in depressed patients. Aust N Z J Psychiatry. 2006 Mar;40(3):225-9. doi: 10.1080/j.1440-1614.2006.01778.x. PMID 16476149
- [Background] Hankin BL, Barrocas AL, Young JF, Haberstick B, Smolen A. 5-HTTLPR x interpersonal stress interaction and nonsuicidal self-injury in general community sample of youth. Psychiatry Res. 2015 Feb 28;225(3):609-12. doi: 10.1016/j.psychres.2014.11.037. Epub 2014 Dec 3. PMID 25500344
- [Background] Gao Y, Xiong Y, Liu X, Wang H. The Effects of Childhood Maltreatment on Non-Suicidal Self-Injury in Male Adolescents: The Moderating Roles of the Monoamine Oxidase A (MAOA) Gene and the Catechol-O-Methyltransferase (COMT) Gene. Int J Environ Res Public Health. 2021 Mar 5;18(5):2598. doi: 10.3390/ijerph18052598. PMID 33807669
- [Background] Strawbridge RJ, Ward J, Ferguson A, Graham N, Shaw RJ, Cullen B, Pearsall R, Lyall LM, Johnston KJA, Niedzwiedz CL, Pell JP, Mackay D, Martin JL, Lyall DM, Bailey MES, Smith DJ. Identification of novel genome-wide associations for suicidality in UK Biobank, genetic correlation with psychiatric disorders and polygenic association with completed suicide. EBioMedicine. 2019 Mar;41:517-525. doi: 10.1016/j.ebiom.2019.02.005. Epub 2019 Feb 8. PMID 30745170
- [Background] Cheung S, Woo J, Maes MS, Zai CC. Suicide epigenetics, a review of recent progress. J Affect Disord. 2020 Mar 15;265:423-438. doi: 10.1016/j.jad.2020.01.040. Epub 2020 Jan 15. PMID 32090769
- [Background] Kang HJ, Bae KY, Kim SW, Shin IS, Hong YJ, Ahn Y, Jeong MH, Yoon JS, Kim JM. BDNF Methylation and Suicidal Ideation in Patients with Acute Coronary Syndrome. Psychiatry Investig. 2018 Oct;15(11):1094-1097. doi: 10.30773/pi.2018.09.20. Epub 2018 Nov 2. PMID 30380818
- [Background] Kang HJ, Kim JM, Lee JY, Kim SY, Bae KY, Kim SW, Shin IS, Kim HR, Shin MG, Yoon JS. BDNF promoter methylation and suicidal behavior in depressive patients. J Affect Disord. 2013 Nov;151(2):679-685. doi: 10.1016/j.jad.2013.08.001. Epub 2013 Aug 13. PMID 23992681
- [Background] Kim JM, Kang HJ, Bae KY, Kim SW, Shin IS, Kim HR, Shin MG, Yoon JS. Association of BDNF promoter methylation and genotype with suicidal ideation in elderly Koreans. Am J Geriatr Psychiatry. 2014 Oct;22(10):989-96. doi: 10.1016/j.jagp.2014.02.011. Epub 2014 Mar 4. PMID 24731781
- [Background] Kim JM, Kang HJ, Kim SY, Kim SW, Shin IS, Kim HR, Park MH, Shin MG, Yoon JH, Yoon JS. BDNF promoter methylation associated with suicidal ideation in patients with breast cancer. Int J Psychiatry Med. 2015;49(1):75-94. doi: 10.1177/0091217415574439. PMID 25838322
- [Background] Zhang Y, Chang Z, Chen J, Ling Y, Liu X, Feng Z, Chen C, Xia M, Zhao X, Ying W, Qing X, Li G, Zhang C. Methylation of the tryptophan hydroxylase-2 gene is associated with mRNA expression in patients with major depression with suicide attempts. Mol Med Rep. 2015 Aug;12(2):3184-90. doi: 10.3892/mmr.2015.3748. Epub 2015 May 7. PMID 25955598
- [Background] Martin-Blanco A, Ferrer M, Soler J, Salazar J, Vega D, Andion O, Sanchez-Mora C, Arranz MJ, Ribases M, Feliu-Soler A, Perez V, Pascual JC. Association between methylation of the glucocorticoid receptor gene, childhood maltreatment, and clinical severity in borderline personality disorder. J Psychiatr Res. 2014 Oct;57:34-40. doi: 10.1016/j.jpsychires.2014.06.011. Epub 2014 Jul 1. PMID 25048180
- [Background] Wang L, Zheng D, Liu L, Zhong G, Bi X, Hu S, Wang M, Qiao D. Relationship between SIRT1 gene and adolescent depressive disorder with nonsuicidal self-injury behavior: Based on gene methylation and mRNA expression. Medicine (Baltimore). 2021 Aug 6;100(31):e26747. doi: 10.1097/MD.0000000000026747. PMID 34397817
- [Background] Zheng D, Bi X, Zhang T, Han C, Ma T, Wang L, Sun M, Cui K, Yang L, Liu L. Epigenetic Alterations of the Promoter Region of the POMC Gene in Adolescent Depressive Disorder Patients with Nonsuicidal Self-injury Behaviors. Psychol Res Behav Manag. 2020 Nov 16;13:997-1008. doi: 10.2147/PRBM.S272445. eCollection 2020. PMID 33235529
- [Background] Mirkovic B, Labelle R, Guile JM, Belloncle V, Bodeau N, Knafo A, Condat A, Bapt-Cazalets N, Marguet C, Breton JJ, Cohen D, Gerardin P. Coping skills among adolescent suicide attempters: results of a multisite study. Can J Psychiatry. 2015 Feb;60(2 Suppl 1):S37-45. PMID 25886670
- [Background] McGirr A, Renaud J, Bureau A, Seguin M, Lesage A, Turecki G. Impulsive-aggressive behaviours and completed suicide across the life cycle: a predisposition for younger age of suicide. Psychol Med. 2008 Mar;38(3):407-17. doi: 10.1017/S0033291707001419. Epub 2007 Sep 6. PMID 17803833
- [Background] Melhem NM, Brent DA, Ziegler M, Iyengar S, Kolko D, Oquendo M, Birmaher B, Burke A, Zelazny J, Stanley B, Mann JJ. Familial pathways to early-onset suicidal behavior: familial and individual antecedents of suicidal behavior. Am J Psychiatry. 2007 Sep;164(9):1364-70. doi: 10.1176/appi.ajp.2007.06091522. PMID 17728421
- [Background] Brodsky BS, Mann JJ, Stanley B, Tin A, Oquendo M, Birmaher B, Greenhill L, Kolko D, Zelazny J, Burke AK, Melhem NM, Brent D. Familial transmission of suicidal behavior: factors mediating the relationship between childhood abuse and offspring suicide attempts. J Clin Psychiatry. 2008 Apr;69(4):584-96. doi: 10.4088/jcp.v69n0410. PMID 18373384
- [Background] Castellvi P, Miranda-Mendizabal A, Pares-Badell O, Almenara J, Alonso I, Blasco MJ, Cebria A, Gabilondo A, Gili M, Lagares C, Piqueras JA, Roca M, Rodriguez-Marin J, Rodriguez-Jimenez T, Soto-Sanz V, Alonso J. Exposure to violence, a risk for suicide in youths and young adults. A meta-analysis of longitudinal studies. Acta Psychiatr Scand. 2017 Mar;135(3):195-211. doi: 10.1111/acps.12679. Epub 2016 Dec 20. PMID 27995627
- [Background] Fergusson DM, Boden JM, Horwood LJ. Exposure to childhood sexual and physical abuse and adjustment in early adulthood. Child Abuse Negl. 2008 Jun;32(6):607-19. doi: 10.1016/j.chiabu.2006.12.018. Epub 2008 Jun 18. PMID 18565580
- [Background] Serafini G, Canepa G, Adavastro G, Nebbia J, Belvederi Murri M, Erbuto D, Pocai B, Fiorillo A, Pompili M, Flouri E, Amore M. The Relationship between Childhood Maltreatment and Non-Suicidal Self-Injury: A Systematic Review. Front Psychiatry. 2017 Aug 24;8:149. doi: 10.3389/fpsyt.2017.00149. eCollection 2017. PMID 28970807
- [Background] Klomek AB, Kleinman M, Altschuler E, Marrocco F, Amakawa L, Gould MS. Suicidal adolescents' experiences with bullying perpetration and victimization during high school as risk factors for later depression and suicidality. J Adolesc Health. 2013 Jul;53(1 Suppl):S37-42. doi: 10.1016/j.jadohealth.2012.12.008. PMID 23790199
- [Background] Kärnä, A., M. Voeten, E. Poskiparta, and C. Salmivalli. 2010. Vulnerable children in varying classroom contexts: Bystanders' behaviors moderate the effects of risk factors on victimization. Merrill-Palmer Quarterly 56:261-82.
- [Background] Hinduja S, Patchin JW. Bullying, cyberbullying, and suicide. Arch Suicide Res. 2010;14(3):206-21. doi: 10.1080/13811118.2010.494133. PMID 20658375
- [Background] Gould MS, Petrie K, Kleinman MH, Wallenstein S. Clustering of attempted suicide: New Zealand national data. Int J Epidemiol. 1994 Dec;23(6):1185-9. doi: 10.1093/ije/23.6.1185. PMID 7721521
- [Background] Gould MS, Wallenstein S, Kleinman M. Time-space clustering of teenage suicide. Am J Epidemiol. 1990 Jan;131(1):71-8. doi: 10.1093/oxfordjournals.aje.a115487. PMID 2293755
- [Background] Fergusson DM, Beautrais AL, Horwood LJ. Vulnerability and resiliency to suicidal behaviours in young people. Psychol Med. 2003 Jan;33(1):61-73. doi: 10.1017/s0033291702006748. PMID 12537037
- [Background] Luthar SS, Cicchetti D, Becker B. The construct of resilience: a critical evaluation and guidelines for future work. Child Dev. 2000 May-Jun;71(3):543-62. doi: 10.1111/1467-8624.00164. PMID 10953923
- [Background] Masten AS, Powell JL. A resilience framework for research, policy, and practice. In: Luthar SS, ed. Resilience and vulnerability: Adaptation in the context of childhood adversities Cambridge: Cambridge University Press; 2003:1-25.
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Whitlock J, Exner-Cortens D, Purington A. Assessment of nonsuicidal self-injury: development and initial validation of the Non-Suicidal Self-Injury-Assessment Tool (NSSI-AT). Psychol Assess. 2014 Sep;26(3):935-46. doi: 10.1037/a0036611. Epub 2014 Apr 21. PMID 24749754
- [Background] Fraley RC, Waller NG, Brennan KA. An item response theory analysis of self-report measures of adult attachment. J Pers Soc Psychol. 2000 Feb;78(2):350-65. doi: 10.1037//0022-3514.78.2.350. PMID 10707340
- [Background] Turin A, Dovc K, Klemencic S, Bratina N, Battelino T, Lipovsek JK, Ursic K, Shmueli-Goetz Y, Drobnic-Radobuljac M. Carer's Attachment Anxiety, Stressful Life-Events and the Risk of Childhood-Onset Type 1 Diabetes. Front Psychiatry. 2021 May 25;12:657982. doi: 10.3389/fpsyt.2021.657982. eCollection 2021. PMID 34140900
- [Background] Dutch SG, Patil N. Validating a Measurement Tool to Predict Aggressive Behavior in Hospitalized Youth. J Am Psychiatr Nurses Assoc. 2019 Sep/Oct;25(5):396-404. doi: 10.1177/1078390318809411. Epub 2018 Dec 20. PMID 30569806
- [Background] Weekers LC, Hutsebaut J, Kamphuis JH. The Level of Personality Functioning Scale-Brief Form 2.0: Update of a brief instrument for assessing level of personality functioning. Personal Ment Health. 2019 Feb;13(1):3-14. doi: 10.1002/pmh.1434. Epub 2018 Sep 19. PMID 30230242
- [Background] Greenwald, R., & Rubin, A. (1999). Assessment of Posttraumatic Symptoms in Children: Development and Preliminary Validation of Parent and Child Scales. Research on Social Work Practice, 9(1), 61-75. https://doi.org/10.1177/104973159900900105
- [Background] Ursic K, Bucik V, Klemencic S, Bratina N, Battelino T, Dovc K, Drobnic Radobuljac M. Validation of the Lifetime Incidence of Traumatic Events (LITE-S/P) Questionnaires in Children and Adolescents in Slovenia. Front Psychiatry. 2021 Jul 1;12:665315. doi: 10.3389/fpsyt.2021.665315. eCollection 2021. PMID 34276439
- [Background] Sharp C, Steinberg L, Temple J, Newlin E. An 11-item measure to assess borderline traits in adolescents: refinement of the BPFSC using IRT. Personal Disord. 2014 Jan;5(1):70-8. doi: 10.1037/per0000057. PMID 24588063
- [Background] Glenn CR, Klonsky ED. One-year test-retest reliability of the Inventory of Statements about Self-Injury (ISAS). Assessment. 2011 Sep;18(3):375-8. doi: 10.1177/1073191111411669. Epub 2011 Jun 10. PMID 21665881
- [Background] Wick RR, Judd LM, Holt KE. Performance of neural network basecalling tools for Oxford Nanopore sequencing. Genome Biol. 2019 Jun 24;20(1):129. doi: 10.1186/s13059-019-1727-y. PMID 31234903
- [Background] Mitsuhashi S, Frith MC, Mizuguchi T, Miyatake S, Toyota T, Adachi H, Oma Y, Kino Y, Mitsuhashi H, Matsumoto N. Tandem-genotypes: robust detection of tandem repeat expansions from long DNA reads. Genome Biol. 2019 Mar 19;20(1):58. doi: 10.1186/s13059-019-1667-6. PMID 30890163
- [Background] Giesselmann P, Brandl B, Raimondeau E, Bowen R, Rohrandt C, Tandon R, Kretzmer H, Assum G, Galonska C, Siebert R, Ammerpohl O, Heron A, Schneider SA, Ladewig J, Koch P, Schuldt BM, Graham JE, Meissner A, Muller FJ. Analysis of short tandem repeat expansions and their methylation state with nanopore sequencing. Nat Biotechnol. 2019 Dec;37(12):1478-1481. doi: 10.1038/s41587-019-0293-x. Epub 2019 Nov 18. PMID 31740840
- [Background] Yuen ZW, Srivastava A, Daniel R, McNevin D, Jack C, Eyras E. Systematic benchmarking of tools for CpG methylation detection from nanopore sequencing. Nat Commun. 2021 Jun 8;12(1):3438. doi: 10.1038/s41467-021-23778-6. PMID 34103501

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT05765864/Prot_SAP_001.pdf